CLINICAL TRIAL: NCT05827887
Title: ProspeCtive Observational Real-world Study of uBRogepant and Atogepant in Israel (COBRA)
Brief Title: An Observational Study to Assess Ubrogepant Tablets and Atogepant Tablets to Treat Migraine in Adult Participants
Acronym: COBRA
Status: Active, not recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P24-078
Record Dates: First submitted 2023-04-13; First posted 2023-04-25 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Migraine
Keywords: Migraine; Ubrogepant; Ubrelvy; Atogepant; Qulipta
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Ubrogepant: Participants will receive ubrogepant as prescribed by their physician in routine clinical practice.
- Atogepant: Participants will receive atogepant as prescribed by their physician in routine clinical practice.

SUMMARY:
Migraine is a neurological disease characterized by moderate or severe headache, associated with nausea, vomiting, and/or sensitivity to light and sound. This study will evaluate how effective the use of ubrogepant and atogepant is in treating adult participants with migraine.

Urogepant (Ubrelvy) and Atogepant (Qulipta) are approved drugs for treatment of migraine in adults in the US. Approximately 200 adult participants who are prescribed Ubrogepant or atogepant by their doctors will be enrolled in this study in Israel.

Participants will receive ubrogepant oral tablets or atogepant oral tablets as prescribed by their physician. Participants will be followed for 90 days.

There is expected to be no additional burden for participants in this trial. Participants will attend regular visits during the study at a hospital or clinic according to their routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of migraine according to the ICHD-3 upon judgement of the treating physician
* The patients should be naive to the designated treatment
* Ability to fill an e-diary app

Exclusion Criteria:

* Patients who cannot be treated with UBRO or ATO according to the applicable approved label
* Patients participating in a concurrent clinical interventional study or within the last 30 days
* Patients who were previously treated with rimegepant will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with migraine prescribed Ubrogepant or Atogepant by their physician.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-06-25 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Ubrogepant (UBRO) Only: Percentage of Participants with Responder Status of "Extremely Satisfied" or "Satisfied" on a Single Item 7-Point Scale | Baseline to Day 90
  The single item 7-point scale asks the question "Overall, how satisfied are you with Ubrelvy for treatment of your migraine?" to assess change in satisfaction of migraine treatment where 0 = extremely satisfied and 6 = extremely dissatisfied.
Atogepant (ATO) Only: Percentage of Participants with Responder Status of "Extremely Satisfied" or "Satisfied" on a Single Item 7-Point Scale | Baseline to Day 90
  The single item 7-point scale asks the question "Overall, how satisfied are you with Qulipta for treatment of your migraine?" to assess change in satisfaction of migraine treatment where 0 = extremely satisfied, 1 = satisfied and 6 = extremely dissatisfied.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (11):
- Israel (11):
  - Edith Wolfson Medical Center /ID# 269740, Holon, Central District
  - Maccabi Healthcare Services /ID# 254171, Kfar Saba, Central District
  - Meir Medical Center /ID# 254170, Kfar Saba, Central District
  - Shaare Zedek Medical Center /ID# 254169, Jerusalem, Jerusalem
  - ZIV Medical Center /ID# 257360, Safed, Northern District
  - Assuta Ashdod Medical Center /ID# 260020, Ashdod, Southern District
  - Soroka University Medical Center /ID# 254551, Beersheba, Southern District
  - The Chaim Sheba Medical Center /ID# 254550, Ramat Gan, Tel Aviv
  - Tel Aviv Sourasky Medical Center /ID# 263089, Tel Aviv, Tel Aviv
  - Clalit HMO /ID# 257364, Gani Tikva
  - Hadassah Medical Center-Hebrew University /ID# 257352, Jerusalem

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=P24-078